CLINICAL TRIAL: NCT03301727
Title: A Pilot Randomized Controlled Trial of Cognitive Behavioural Therapy for Insomnia in Pregnancy
Brief Title: Sleeping for Two: RCT of CBT-Insomnia in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB15-2137
Record Dates: First submitted 2017-09-22; First posted 2017-10-04 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2017-09

CONDITIONS: Insomnia; Sleep Disturbance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- In-person CBT-I Treatment (Active Comparator): Participants receive 6 in-person weekly 1.5-hour sessions of cognitive-behavioural therapy for insomnia (CBT-I) for pregnant women, supervised by a registered, licensed clinical psychologist.
  Interventions: Other: Cognitive-Behavioural Therapy for Insomnia (CBT-I)
- Online CBT-I Treatment (Active Comparator): Participants receive 6 online weekly 1.5-hour sessions of cognitive-behavioural therapy for insomnia (CBT-I) for pregnant women, supervised by a registered, licensed clinical psychologist.
  Interventions: Other: Cognitive-Behavioural Therapy for Insomnia (CBT-I)
- Wait-list Control (Other): Participants are placed on a wait-list for 6 weeks before receiving either in-person or online 6 weekly 1.5-hour sessions of cognitive-behavioural therapy for insomnia (CBT-I) for pregnant women, supervised by a registered, licensed clinical psychologist.
  Interventions: Other: Cognitive-Behavioural Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Other: Cognitive-Behavioural Therapy for Insomnia (CBT-I) — Cognitive-Behavioural Therapy for Insomnia (CBT-I) is an evidence-based psycho-therapeutic intervention, combining cognitive and behavioural principles to provide psycho-education concerning contributing thoughts to sleep problem maintenance, and behavioural technique instruction to reduce sleep onset latency and promote effective sleep maintenance.
  Other Names: Cognitive-Behavioral Therapy for Insomnia (CBT-I)

SUMMARY:
Cognitive-behavioural therapy for insomnia (CBT-I) has been shown to be an effective treatment for insomnia in multiple populations, including women during pregnancy and postpartum. Online CBT-I has also been shown to be effective and comparable to in-person CBT-I, and shows promise as an accessible treatment alternative to in-person CBT-I for pregnant women experiencing insomnia. As the harmful consequences of insomnia or sleep disturbances have been well documented during late pregnancy, this randomized-controlled trial will compare the efficacy of both in-person and online CBT-I on pregnant women with insomnia to a wait-list control group.

DETAILED DESCRIPTION:
The primary aim of the current project is to evaluate the impact of a 6-week in-person CBT-I, versus online CBT-I, versus a wait-list in reducing symptoms of insomnia (assessed subjectively by self-report and objectively with actigraphy) experienced in pregnancy. The investigators hypothesize that participants who receive a 6-week program of either in-person CBT-I or online CBT-I (versus a wait-list) will report fewer insomnia symptoms and have improved objectively assessed sleep measured at one-week post-treatment. Based on previous research findings, the investigators do not expect that there will be a difference between in-person CBT-I and online CBT-I administration.

The secondary aim is to investigate if CBT-I versus a wait-list will reduce symptoms of depression at one-week post-treatment. The investigators hypothesize that participants who receive in-person CBT-I and online CBT-I (versus a wait-list) will report fewer depressive symptoms measured at one-week post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or greater
* Gestation: 12 - 30 weeks
* Identifying as experiencing sleep disturbances
* Language: English-intermediate or above
* Have access to internet

Exclusion Criteria:

* Experiencing symptoms of sleep disorders other than insomnia
* Currently taking prescribed medications for sleep problems
* History of untreated, serious psychiatric illness
* Substance-use during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in the Insomnia Severity Index | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  The ISI is a 7-item questionnaire designed to identify cases of insomnia and evaluate treatment outcomes. The ISI assesses severity of sleep onset, sleep maintenance and early wakening problems, sleep dissatisfaction, and perceived distress caused by sleep problems. It was found to be a clinically useful tool in assessing changes in insomnia symptoms in insomnia treatment research.
Change in the Pittsburgh Sleep Quality Index | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  The PSQI instrument is used in assessing one's sleep quality during the previous month. It consists of 19 self-rated items and 5 questions rated by the roommate or bed partner. There are seven components of the PSQI and these are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction.
Change in Actigraphy (Actiwatch II, Phillips, USA) | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  Actigraphy monitoring provides objective sleep, combining measurements of: circadian rhythm amplitude, acrophase, mesor, sleep efficiency, sleep latency, total sleep time, and number and frequency of awakenings.
Change in Sleep Logs | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  Sleep logs provide self-reported subjective sleep, combining self-reports of: latency, total sleep time, and number and frequency of awakenings.

SECONDARY OUTCOMES:
Change in the Edinburgh Postpartum Depression Scale | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  Symptoms of depression in pregnancy and the postpartum will be assessed by the EPDS. The EPDS consists of 10 items and is a reliable and valid tool for identifying symptoms of depression experienced in pregnancy and the postpartum.

OTHER OUTCOMES:
Change in the Multidimensional Fatigue Symptom Inventory - Short Form | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  30-item short form version of MFSI was designed to assess manifestations of fatigue.
Change in the Dysfunctional Beliefs and Attitudes about Sleep Questionnaire | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  Cognitive scale of 16 items used for assessing problematic levels of unhelpful beliefs about sleep.
Change in the Sleep Self-Efficacy Scale | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  9-item scale used for measuring one's level of confidence in carrying out specific sleep-related behaviors.
Change in the Sleep Hygiene Index | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  13-item self-report items used for assessing presence of behaviors thought to compromise sleep hygiene.
Change in the Pre-Sleep Arousal Scale | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  16-item self-report measure assessing pre-sleep arousal.
Change in the Glasgow Sleep Effort Scale | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  Measure of sleep-related effort.
Change in the Sleep-Related Behaviors Questionnaire | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  Designed to assess use of safety behaviours to promote sleep and cope with tiredness.
Change in the Epworth Sleepiness Scale | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  8-item scale designed to assess the tendency to fall asleep in situations
Change in the Generalized Anxiety Disorder index | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  Brief measure for assessing symptoms of generalized anxiety disorder.
Change in the Couple Satisfaction Index | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  16-item scale assessing participants' relationship satisfaction.
Change in the Big Five Inventory | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  44-items assessing personality.
Change in the Extended Brief Infant Sleep Questionnaire | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  24-items assessing infant sleep.
Change in the Pregnancy-Specific Anxiety Measure | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  4-items assessing anxiety during pregnancy.
Change in the PROMIS Adult Version 1.0 Pain Interference Short Form 8a | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  8-items assessing interference of pain in functioning.
Change in the PROMIS Adult Version 1.0 Pain Intensity Short Form 3a | Change between 3 time-points: baseline, 8-week follow-up, 3-months postpartum follow-up
  3-items assessing intensity of pain symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Lianne Tomfohr-Madsen, PhD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba

REFERENCES:
- [Derived] MacKinnon AL, Silang K, Watts D, Kaur J, Freeman M, Dewsnap K, Keys E, Madsen JW, Giesbrecht GF, Williamson T, Metcalfe A, Campbell T, Mrklas KJ, Tomfohr-Madsen LM. Sleeping for Two: a randomized controlled trial of cognitive behavioral therapy for insomnia in pregnancy. J Clin Sleep Med. 2025 Feb 1;21(2):365-376. doi: 10.5664/jcsm.11396. PMID 39436396

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT03301727/Prot_SAP_000.pdf